CLINICAL TRIAL: NCT06553794
Title: Protein Digestion and Amino Acid Absorption in the Aging Gastrointestinal Tract
Acronym: AgingGut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: METC23-029
Record Dates: First submitted 2023-06-27; First posted 2024-08-14 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Protein Malabsorption
Keywords: Protein; Digestion; Absorption; Intestinal mucosa; Aging
MeSH Terms: interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Non-therapeutic intervention (Experimental): Subjects will undergo a standardized heavy water dosing protocol for 2 days (1 "loading day", 1 "maintenance day") and consume a standardized diet for 2 days. On the experimental test day, a gastroscopy with collection of duodenal mucosa tissue samples will be performed.
  Interventions: Other: Gastroscopy with duodenal mucosal tissue biopsies

INTERVENTIONS:
Other: Gastroscopy with duodenal mucosal tissue biopsies — Subjects will undergo a standardized heavy water dosing protocol for 2 days (1 "loading day", 1 "maintenance day") and consume a standardized diet for 2 days. On the experimental test day, a gastroscopy with collection of duodenal mucosa tissue samples will be performed.

SUMMARY:
Rationale: Worldwide, the aging population is increasing. Aging is associated with loss of independence and increased risk of co-morbidity. Sufficient protein intake is imperative to maintain skeletal muscle mass and overall health, and thereby stimulates active aging. It has been suggested that age-dependent changes in gastrointestinal (GI) tract physiology affect the amount of protein digested and absorbed, as well as the intestinal microbiota. However, it is not clear to what extent actual protein digestion and absorption are altered in older individuals. So far, no human data on the expression and activity of brush border enzymes and protein-related transporters in small intestinal epithelial cells are available. Understanding the age-dependent digestion and absorption kinetics of protein is important for creating specific diets in older individuals to improve protein intake and thereby stimulate healthy aging.

Objective: To assess the effects of aging on protein digestion and amino acid absorption in healthy humans in vivo.

Study design: Cross-sectional Study population: 12 healthy, non-obese (BMI 18.5-30kg/m2) young adults (age: 18-35 y inclusive) and 12 community dwelling older adults (age: ≥67 y).

Intervention: Subjects will undergo a standardized heavy water dosing protocol for 2 days (1 "loading day", 1 "maintenance day"). Blood and saliva sampling will be conducted throughout the heavy water dosing protocol to determine body water and amino acid enrichment levels. On the experimental test day, a gastroscopy with collection of duodenal mucosa tissue samples will be performed to allow assessment of the expression and activity of brush border enzymes and protein-related transporters, and to determine fractional duodenal mucosal protein synthesis rate. Fecal samples will be collected at baseline and after the gastroscopy.

Main study parameters/endpoints: The primary study parameter is the mRNA expression of brush border enzymes and small peptide and amino acid transporters in duodenal mucosal cells. Secondary study parameters include protein expression of brush border enzymes and small peptide and amino acid transporters in duodenal mucosal cells, fecal microbial fermentation metabolites and duodenal mucosal protein synthesis rate.

DETAILED DESCRIPTION:
Worldwide, the proportion of older individuals in the population is increasing. The progressive loss of skeletal muscle mass with aging, or sarcopenia, has a major impact on our health care system and costs due to increased morbidity and a greater need for hospitalization and/or institutionalization. A sufficient protein intake is imperative to maintain skeletal muscle mass and overall health, and thereby stimulates active aging. Whereas the overall protein intake is generally lower in older as compared to young adults, findings indicate that older adults need more protein to increase muscle protein synthesis, known as anabolic resistance. The exact mechanisms underlying anabolic resistance are not fully discovered yet. Age-dependent changes in gastrointestinal tract physiology have been suggested as a potential cause.

Following protein ingestion, protein is cleaved into small peptides and amino acids by digestive enzymes secreted in the stomach (pepsin) and small intestinal lumen (pancreatic trypsin, chymotrypsin, elastase), as well as brush border enzymes (aminopeptidase, carboxypeptidase, dipeptidase). Brush border enzymes are responsible for the final digestion of small peptides into dipeptides, tripeptides and amino acids. Subsequently, these small peptides and amino acids are absorbed across the intestinal mucosa by various membrane-bound transporters. The majority of dietary-protein derived amino acids is released into the systemic circulation and transported and taken up by various peripheral tissues in the postprandial phase.

It has been shown that postprandial plasma amino acid availability is lower in older compared to young adults. This indicates that digestion and absorption of proteins are likely attenuated in older individuals, thereby reducing the systemic availability of protein-derived amino acids for muscle protein synthesis and other relevant physiological processes.

Limited studies have focused on changes in gastrointestinal tract physiology with aging. Human studies on the expression and activity of brush border enzymes and protein transporters (i.e. for dipeptides, tripeptides and amino acids) being crucial for the final steps of digestion and absorption, respectively, are lacking. Therefore, the aim of the present study is to assess the expression and activity of brush border enzymes and expression of protein transporters in small intestinal epithelial cells in older as compared to young adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35 years or 67+ years
* Body mass index (BMI) between 18.5 and 30 kg/m2
* Regular stool frequency ranging from 1-3 times/day

Exclusion Criteria:

* History of cardiovascular, respiratory, gastrointestinal, urogenital, neurological, psychiatric, dermatologic, musculoskeletal, metabolic, endocrine, haematological, immunologic disorders, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol, interfere with the execution of the experiment, or potential influence the study outcomes (to be decided by the principal investigator and responsible physician)
* Major abdominal surgery interfering with gastrointestinal function (upon judgement of the principal investigator and responsible physician)
* Use of medication which limit participation in or completion of the study protocol, interferes with the execution of the experiment, or potential influences the study outcomes (to be decided by the principal investigator and responsible physician)
* Use of supplementation (i.e. protein, vitamin, pre- and probiotic supplementation) within 14 days prior to testing
* Administration of investigational drugs or participation in any scientific intervention study prior or during the study, which may interfere with this study (upon judgement of the principal investigator and responsible physician) Specific diet (e.g. vegetarian, vegan, gluten free, no diary) within the study period
* Planning to lose weight during the study period
* Excessive alcohol consumption (defined as > 14 alcoholic consumptions per week)
* Smoking
* Drug use
* Pregnancy
* Lactation
* Donated blood three months prior to the test day
* No given permission to register participation in electronic patient file at MUMC+ and to add records of gastroduodenoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
Gene expression of brush border enzymes and protein-related transporters in duodenal mucosal cells | day 3 of study period
  as determined by real-time polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
Protein expression of brush border enzymes and protein-related transporters | day 3 of study period
  as determined by proteomic analysis
Microbial proteolytic fermentation metabolites involved in protein metabolism | Baseline
  as determined by high performance liquid chromatography-mass spectrometry
Fractional duodenal mucosal protein synthetic rate | during study period (3 days)
  as determined using stable isotope tracer methodology (D2O)
Fecal elastase | Baseline
  as marker for pancreatic enzyme secretion
Plasma citrulline | Baseline
  as a marker for total functional enterocyte mass

OTHER OUTCOMES:
Age in years | Baseline
  Reported by participants
Body weight in kg | Baseline
  Scale
Height in m | Baseline
  Stadiometer
BMI in kg/m2 | Baseline
  Calculated based on height and weight
Blood pressure in mmHg | Baseline
  Electrical sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Jonkers, Prof, Principal Investigator — Maastricht University Medical Center; Luc van Loon, Prof, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No